CLINICAL TRIAL: NCT06208371
Title: The DECIDE-CRLM-10 Randomized Controlled Study: Comparison of Chemotherapy Combined With Localized Treatment for Liver Metastases Versus Palliative Chemotherapy Alone in Colorectal Patients With 10 or More Liver Metastases
Brief Title: Localized Treatment Versus Palliative Chemotherapy in CRC Patients With 10 or More CRLM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECIDE-CRLM-10
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: Colorectal liver metastases; Overall survival; Locoregional treatment; Palliative chemotherapy; Randomized Clinical Study
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants who meet the inclusion criteria will be grouped using a stratified block randomization method. The stratification factors include the entire RAS/BRAF gene (wild-type vs. mutated), the number of liver metastases (10-20 vs. >20), and the location of the primary lesion (left vs. right). The random grouping of participants will be accomplished using our center's Interactive Web Response System (IWRS). The participants will be randomly assigned to either the liver-localized treatment group or the palliative chemotherapy group in a 2:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liver-localized treatment group (Experimental): Participants in this group will undergo liver-localized interventions, which may include surgical resection and/or ablation therapy and/or SBRT, aiming to achieve NED.
  Interventions: Procedure: Surgical resection and/or ablation therapy and/or SBRT
- Palliative chemotherapy only group (Active Comparator): Participants in this group will receive standard palliative chemotherapy. The focus is on managing symptoms and controlling the progression of the disease.
  Interventions: Drug: Palliative Chemotherapy

INTERVENTIONS:
Procedure: Surgical resection and/or ablation therapy and/or SBRT — Participants may receive surgical resection and/or ablation therapy and/or stereotactic body radiotherapy
  Arms: Liver-localized treatment group
Drug: Palliative Chemotherapy — Participants in this group may continue the original systemic chemotherapy regimen. Patients with tumor control after 10-12 cycles can either transition to maintenance treatment or temporarily suspend treatment until disease progression, at which point they switch to a second-line treatment regimen.The selection of second-line and subsequent treatment regimens follows CSCO guidelines and clinical practices.
  Arms: Palliative chemotherapy only group

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of localized interventions in improving the 5-year survival rate for colorectal cancer patients with ≥10 liver metastases. We aim to answer the following question:

Can localized interventions, including surgery and/or ablation and/or stereotactic body radiotherapy (SBRT), enhance the 5-year survival rate compared to palliative chemotherapy alone in patients with ≥10 colorectal liver metastases (CRLM)?

Participants in this study, who have achieved disease control through chemotherapy, will undergo either localized interventions (surgery and/or ablation and/or SBRT) or receive palliative chemotherapy alone. Researchers will compare the survival outcomes between these groups to determine the potential benefits of localized interventions for patients with ≥10 CRLM.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignant tumors, ranking second globally in cancer-related mortality. In recent years, both the incidence and mortality rates of colorectal cancer in China have shown a gradual upward trend. According to literature reports, 20% of colorectal cancer patients are diagnosed with liver metastases (CRLM), and as the disease progresses, up to 50% of patients may develop liver metastases, a primary cause of treatment failure for these patients. Surgical resection of liver metastases remains the main curative treatment for colorectal cancer patients, with 5-year and 10-year survival rates reaching 33% and 23%, respectively. However, only 15%-20% of patients are eligible for liver surgery. Advances in targeted drugs and systemic chemotherapy in recent years have improved the response rate of colorectal cancer patients with liver metastases. Several clinical studies confirm that neoadjuvant chemotherapy can reduce the size and stage of liver metastases, allowing initially unresectable patients the opportunity for surgical intervention. Simultaneously, various local treatment modalities for colorectal liver metastases, including surgery, ablation therapy, and stereotactic body radiotherapy (SBRT), have evolved, aiming to achieve no evidence of disease (NED).

However, not all patients benefit from liver metastasis surgical resection, and the number of liver metastases is a crucial factor influencing the prognosis of colorectal cancer patients undergoing liver surgery. In the 1970s and 1980s, it was considered a contraindication for surgery if there were more than 3 liver metastatic lesions. In a subsequent phase II clinical trial, the CLOCC study, 119 initially unresectable colorectal cancer patients with fewer than 10 metastatic lesions were randomized into either palliative chemotherapy (control group) or systemic chemotherapy combined with liver ablation ± surgical resection (experimental group). The overall survival of patients in the combination therapy group was significantly higher than that in the palliative chemotherapy group (HR=0.58, 95% CI 0.38-0.88, p=0.01). The 3-year, 5-year, and 8-year survival rates in the combination therapy group were 56.9%, 43.1%, and 35.9%, respectively, confirming that for colorectal cancer patients with fewer than 10 unresectable liver metastases, the efficacy of systemic chemotherapy combined with surgery and ablation therapy is superior to palliative chemotherapy alone.

To explore the impact of surgical resection on the survival of colorectal cancer patients with ≥10 liver metastases after first-line treatment, several retrospective studies have been conducted. A study by L. Viganò et al. found that in 106 colorectal cancer patients with ≥8 metastatic lesions, the 5-year survival rate and 5-year recurrence-free survival rate after surgical resection were 20.1% and 13.6%, respectively. There was no significant difference in the 5-year survival rate among patients with 8-10, 10-15, and ≥15 metastatic lesions (p=0.848). Multifactorial analysis of patients with ≥ 8 metastatic lesions showed that the presence of extrahepatic lesions before surgery (HR=2.38, 95% CI 1.23-4.60, p=0.010) and poor response to preoperative chemotherapy (HR=2.14, 95% CI 1.11-4.12, p=0.023) were independent risk factors for overall survival in patients with ≥10 CRLM. Another large observational study by M. A. Allard included 529 patients with ≥10 liver metastases, yielding an overall 5-year survival rate of 30%. Among the colorectal cancer patients with ≥10 lesions, 68.4% (362/529) received chemotherapy before surgery, and 96.3% of these patients underwent surgical resection when the disease was controlled or stable. 72.8% patients underwent R0 or R1 ± ablation therapy, while 27.2% underwent R2 resection or did not undergo surgical resection. Patients who underwent R0 resection and R1 resection ± ablation therapy had better 3-year and 5-year survival rates than those who underwent R2 resection or did not undergo surgical resection (61% and 39% vs. 29% and 5%; p<0.0001). The study also found that among these patients, there was no significant difference in the 3-year and 5-year survival rates between those who underwent R0 resection and R1 resection ± ablation therapy (73% and 45% vs. 60% and 44%; p<0.72), and those who underwent R2 resection or did not undergo surgical resection (29% and 6% vs. 28% and 0%; p=0.77). The results of this study also showed that among patients with ≥10 CRLM, those who underwent MRI before surgery, achieved R0/R1 resection, and received adjuvant therapy after surgery had a longer survival.

Furthermore, Lin et al. used univariate and multivariate analysis to identify ≥10 liver metastases as an independent prognostic factor for colorectal cancer patients with CRLM (HR=1.629; 95% CI 1.007-2.636; p=0.043). Subsequently, a retrospective study was conducted specifically for colorectal cancer patients with liver metastases using 10 metastases as the cutoff value. The results showed that the conversion rate of patients with ≥10 liver metastases (43.4%) was significantly lower than that of patients with <10 liver metastases (57.3%; p=0.001). Among successfully converted patients, the 2-year survival rate of patients with <10 liver metastases was significantly higher than that of patients with ≥10 liver metastases (89.9% [95% CI 82.5%-98.0%] vs. 58.2% [95% CI 42.2%-80.4%], p=0.008). In patients with ≥10 liver metastases, there was no significant difference in the 2-year survival rate between those who successfully underwent conversion surgery and those who did not (58.2% [95% CI 42.2%-80.4%] vs. 49.6% [95% CI 37.5%-65.7%], p=0.160). For patients with <10 CRLM, the 2-year survival rate of successfully converted patients was significantly higher than that of those who did not convert successfully (89.9% [95% CI 82.5%-98.0%] vs. 58.9% [95% CI 45.2%-76.7%], p<0.001).

In summary, for colorectal cancer patients with liver metastases, adopting a locoregional treatment approach can enhance the survival of those with <10 liver metastatic lesions. However, significant controversy remains regarding whether surgical treatment significantly improves the survival of colorectal cancer patients with ≥10 CRLM. Currently, there is a lack of randomized controlled study data to address the question of whether colorectal cancer patients with ≥10 CRLM can further benefit from chemotherapy plus a surgical approach versus palliative chemotherapy alone.

To that end, the present study will focus on patients with ≥10 CRLM who have achieved disease control in liver metastatic lesions after chemotherapy and can potentially attain a disease-free state through surgery and/or ablation and/or stereotactic body radiotherapy (SBRT). The primary objective of this study is to investigate whether liver-localized intervention can improve the 5-year survival rate compared to palliative chemotherapy, for colorectal cancer patients with ≥10 CRLM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed colorectal adenocarcinoma.
* Baseline imaging (CT, MRI, or PET/CT as necessary) or pathological confirmation of liver metastasis, with no extrahepatic metastasis (consideration for inclusion may be given to lesions with a diameter less than 10mm in the lungs or lymph nodes if metastasis is difficult to confirm or is suspected).
* Disease control (PR or SD) achieved after a minimum of 8 cycles of systemic chemotherapy.
* Evaluation by a centralized liver surgeon expert group to confirm presence of ≥10 liver metastases, which can be managed through surgery and/or ablation and/or SBRT to achieve NED. Non-resectability is defined as one or more of the following: ① Unable to undergo R0 resection; ② Predicted insufficient remaining liver volume after resection; ③ After resection, none of the three hepatic veins can be preserved, and the preservation of residual liver inflow and outflow and bile ducts cannot be guaranteed, and adjacent two liver segments cannot be preserved.
* Curative surgery possible for the primary colorectal lesion.
* Normal hematological, hepatic, and renal functions at baseline.
* Child-Pugh grade A liver function.
* ECOG performance status 0-1.
* Tolerability to undergo further surgery and chemotherapy.
* Life expectancy > 3 months.
* Signed written informed consent.
* Willing and able to undergo follow-up until death, study completion, or study termination.

Exclusion Criteria:

* Definite presence of extrahepatic metastasis and/or primary tumor not amenable to curative surgical resection.
* Severe arterial embolism or ascites.
* Bleeding tendencies or coagulation disorders.
* Hypertensive crisis or hypertensive encephalopathy.
* Severe uncontrollable systemic complications such as infection or diabetes.
* Clinically severe cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), uncontrolled hypertension despite appropriate medical treatment, unstable angina, congestive heart failure (NYHA 2-4), and arrhythmias requiring medication.
* History or physical examination indicating central nervous system diseases (such as primary brain tumor, uncontrollable epilepsy, any brain metastasis, or history of stroke).
* Diagnosis of other malignant tumors within the past 5 years (excluding basal cell carcinoma after radical surgery and/or cervical carcinoma in situ).
* Pregnant or lactating women.
* Women of childbearing potential not using or refusing to use effective non-hormonal contraceptive methods (intrauterine devices, combined barrier contraceptive methods with spermicidal gel, or sterilization) or men with reproductive potential.
* Inability or unwillingness to comply with the study protocol.
* Any other diseases, metastatic lesions causing functional impairment, or suspicious findings in the physical examination indicating possible contraindications for the use of investigational drugs or placing the patient at a high risk of treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Five-year survival rate | Assessed five-year following diagnosis
  The proportion of patients who are still alive five years following diagnosis

SECONDARY OUTCOMES:
Median Progression-Free Survival | Assessed throughout the study duration (5 years)
  The duration of time from the initiation of treatments until disease progression or death.
Median Overall Survival | Assessed throughout the study duration (5 years)
  The duration of time from diagnosis until death
Cumulative Incidence of Liver Progression Events | Assessed throughout the study duration (5 years)
  The proportion of patients experiencing disease progression specifically in the liver over the study period.
Cumulative Incidence of Extrahepatic Progression Events | Assessed throughout the study duration (5 years)
  The proportion of patients experiencing disease progression outside the liver over the study period.
Treatment-related Adverse Events | Assessed throughout the study duration (5 years)
  Assessment of adverse events related to surgical interventions, including but not limited to complications compared to palliative chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.